CLINICAL TRIAL: NCT02108535
Title: Comparative Analysis of Cost-effectiveness of Silver Dressing in Burns
Acronym: ARGENTUM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sorocaba (Other)
Responsible Party: Principal Investigator, Luciane Cruz Lopes, Professor - Researcher, University of Sorocaba
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UNISO-2012
Record Dates: First submitted 2014-04-05; First posted 2014-04-09 (Estimated); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Second-degree Burn
Keywords: burns; dressings; silver sulfadiazine; silver compounds; cost
MeSH Terms: conditions — Burns | interventions — Acticoat; Silver Sulfadiazine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nanocrystalline silver (Experimental): Flexible polyester low-grip coated nanocrystalline silver dressing. The dressing was applied to the lesion after being soaked in sterile distilled water. About this compresses to bandage movements will have been added and comes to avoid tourniquet bandage on-site maintenance, temperature of the affected area, cushioning and absorption of wound exudate when present. Is finished with the application of crepe bandages in the form of flakes containment curative and maintenance of pressure. This procedure aids in the bloodstream, and avoids the increased edema. The bandage is started from the periphery to the central region, avoiding tourniquet. The exchanges were performed every three days.
  Interventions: Drug: Nanocrystalline silver
- Silver sulfadiazine (Active Comparator): Ranges for rayon containing cream 1% silver sulfadiazine were used. Involving this layer, bandages for dressings were added in movements back and forth to avoid the tourniquet, providing maintenance of the temperature of the affected area, cushioning and absorption of wound exudate when present. This application was completed with crepe bandages to contain the dressing and maintain pressure. This procedure aids in the bloodstream, and avoids the increased edema. The bandage is started from the periphery to the central region, scales, avoiding the tourniquet. Dressing changes were performed daily.
  Interventions: Drug: Silver Sulfadiazine

INTERVENTIONS:
Drug: Nanocrystalline silver — Flexible polyester low-grip coated nano-crystalline silver layer. The level of silver is 1.64 mg/ cm². This dressing enables the sustained release of silver in humid conditions dynamically and reached a higher plateau than 60 mg / L in less than 2 hours, and maintains a uniform level by 72 hours.
  Other Names: Acticoat
  Arms: Nanocrystalline silver
Drug: Silver Sulfadiazine — This is at Standard treatment. The cream silver sulphadiazine at 1% was applied on the burn aseptically in a thick layer, approximately 3 to 5 mm, ie 5 g per 80 cm2
  Other Names: Silvazine
  Arms: Silver sulfadiazine

SUMMARY:
The evidence is insufficient to determine whether the types of dressings containing silver differ in time / proportion for complete wound healing and pain. We will analyze the cost-effectiveness of these dressings in outpatients, considering the service provided by the Brazilian National Public Health System.

DETAILED DESCRIPTION:
Randomized, single-center, single-blinded, controlled clinical trial. Adult patients (age between 18 and 65 years), regardless of sex, with second degree burns treated in outpatient regimen will be randomized (1:1) into two groups: 1% silver sulfadiazine and nanocrystalline silver.

Primary outcome:

- Proportion of lesions completely epithelialized within 15 days.

Secondary outcomes:

* Time in days for complete epithelialization of the burned areas;
* Number of dressing changes;
* Level of pain associated with the application and removal of the dressings;
* Direct medical and non-medical costs;
* Need for surgery;
* Incidence of infection;
* Presence of local adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18 and 65 years;
* Regardless of sex and ethnicity;
* Presenting second degree burns (partial thickness involving the epidermis and part of the dermis, with at least the preservation of some dermal appendages from of which the wound can eventually be epithelialized spontaneously) (ARTZ; MONCRIEF; PRITT, 1980) under an outpatient regimen, without the need for surgical debridement of devitalized tissue and skin grafts informed in the initial clinical diagnosis.

Exclusion Criteria:

* Patients with diabetes;
* Pregnant women;
* Patients with intellectual disabilities;
* Patients with burns to the face or on the palmar face of the hands or on the plantar face of the feet, as the need for specific treatment was felt to prevent functional sequelae;
* Patients who have already started treatment in other institutions;
* Those whose burns had happened 5 or more days before their entrance in the hospital;
* Those incapable of signing the informed consent form or who have declined to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-11; Primary Completion 2014-08 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Complete epithelialization of the wound | 15 days
  Proportion of lesions completely epithelialized during the specific time frame

SECONDARY OUTCOMES:
Number of dressing changes | 30 days
  The number of dressing changes in the patients
Direct medical and non-medical costs of treatment | 15 days
  The medical and non-medical cost of the treatment comparing both dressings
Level of pain | 30 days
  Level of pain associated with the application and removal of dressings
Sugery | 90 days
  The need for surgery
Infection | 30 days
  The incidence of infection
Adverse reactions | 90 days
  Any adverse reactions caused by the silver dressings

CONTACTS AND LOCATIONS:
Overall Officials: Luciane C Lopes, PhD, Principal Investigator — UNISO
Locations (1):
- Clinic of the Burn Treatment of Sorocaba's Hospital Complex, Sorocaba, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moreira SS, Camargo MC, Caetano R, Alves MR, Itria A, Pereira TV, Lopes LC. Efficacy and costs of nanocrystalline silver dressings versus 1% silver sulfadiazine dressings to treat burns in adults in the outpatient setting: A randomized clinical trial. Burns. 2022 May;48(3):568-576. doi: 10.1016/j.burns.2021.05.014. Epub 2021 Jun 1. PMID 34688520